CLINICAL TRIAL: NCT06750029
Title: How Does Medical Clown Intervention Affect the Length of Hospitalization in Children With Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Karin Yaakobi Bianu, Medical Doctor, Carmel Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMC-0170-16
Record Dates: First submitted 2024-12-06; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Community-Acquired Pneumonia (CAP)
Keywords: Medical clowns; Community-Acquired Pneumonia (CAP)
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigation Group (Experimental): Investigation group will be receiving standard care plus 15-minute MC visits twice daily during the first 48 hours of hospitalization
  Interventions: Other: Medical clown visits
- Control Group (No Intervention): Control Group will be receiving standard care without MC visits.

INTERVENTIONS:
Other: Medical clown visits — The intervention is 15-minute visits from MCs twice daily during the first two days of admission. The clowns use various techniques to relax the patients (e.g. music, singing, playing, humor, guided imagination) and helpe encourage children to begin drinking and eating on their own.
  Other Names: Medical Clown
  Arms: Investigation Group

SUMMARY:
Background and Objectives: Community-acquired pneumonia (CAP) is a leading cause of hospitalization in children. The hospitalization duration depends on factors as child's well-being, vital signs, need for parenteral treatments, and development of complications. Medical clowns (MCs) are known to assist in reducing pain and alleviating anxiety and have been integrated into many aspects of hospital treatment routines. The aim of this study is to evaluate the effect of MC intervention on length of hospitalization in children admitted with CAP.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of pneumonia.
* Ages 2-18 years.

Exclusion Criteria:

* Hemodynamically unstable patients.
* Other systemic comorbidities or chronic respiratory diseases
* Children from families unable to comprehend and sign an informed consent form.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
The length of hospitalization in hours | Immediately after the intervention
  The length of hospitalization in hours is determined by the duration between admission and discharge from the pediatric department.

SECONDARY OUTCOMES:
Duration of IV treatment | Immediately after the intervention
  Duration of IV treatment in hours.

OTHER OUTCOMES:
Changes in well-being scores as reported by both the parent and the treating physician. | Immediately after the intervention
  Changes in well-being scores as reported by both the parent and the treating physician, and alterations in vital signs and laboratory results.
Alterations in Heart rate | Immediately after the intervention
  Alterations in Heart rate
Alterations in body temperature | Immediately after the intervention
  Alterations in body temperature
Alterations in Respiratory rate | Immediately after the intervention
  Alterations in Respiratory rate
Alterations in oxygen saturation | Immediately after the intervention
  Alterations in oxygen saturation
Alterations in white blood cell count | Immediately after the intervention
  Alterations in white blood cell count
Alterations in absolute neutrophil count | Immediately after the intervention
  Alterations in absolute neutrophil count
Alterations in C-reactive protein levels | Immediately after the intervention
  Alterations in C-reactive protein levels

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khoury L, Shwartz Naddam I, Paz Tzruia M, Shehadeh S, Konopnicki M, Hamad Saied M, Meiri N, Livnat G, Yaacoby-Bianu K. Medical clown intervention shortens length of hospitalization in children with pneumonia. Sci Rep. 2025 Jun 4;15(1):19498. doi: 10.1038/s41598-025-04706-w. PMID 40461561

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT06750029/Prot_SAP_000.pdf